CLINICAL TRIAL: NCT02309840
Title: The Modifying Eating and Lifestyles at School (MEALS) Study
Brief Title: The Modifying Eating and Lifestyles at School Study
Acronym: MEALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Eric B. Rimm, Professor of Epidemiology and Nutrition, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 21198-103
Record Dates: First submitted 2014-11-18; First posted 2014-12-05 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Meals; Food Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control (No Intervention): Students received standard meals in a standard cafeteria environment
- Chef (Experimental): Students were exposed to chef-enhanced meals
  Interventions: Other: Chef-enhanced meals
- choice architecture (Experimental): Students were exposed to modifications to the physical environment in the cafeteria to "nudge" students towards healthier choices
  Interventions: Behavioral: choice architecture
- Chef and choice architecture (Experimental): Students were exposed to both chef-enhanced meals and modifications to the physical environment in the cafeteria to "nudge" students towards healthier choices
  Interventions: Behavioral: choice architecture; Other: Chef-enhanced meals

INTERVENTIONS:
Behavioral: choice architecture — 1. Place vegetables at the beginning of the lunch line.
  2. Place fruits in attractive bowls or trays lined with appealing fabric, and place other fruit options next to the cash registers.
  3. Promote fruits and vegetables with prominently displayed signage and images.
  4. Place white milk selection in front of sugar-sweetened milk (e.g. chocolate milk) or at eye-level.
  Other Names: Smart Cafe
  Arms: Chef and choice architecture; choice architecture
Other: Chef-enhanced meals — meals prepared by a professional chef with enhanced palatability
  Arms: Chef; Chef and choice architecture

SUMMARY:
The purpose of this study is to examine the impact of introducing healthier, chef-enhanced foods and/or environmental modifications (choice architecture) on selection and consumption of school foods among elementary and middle school students.

DETAILED DESCRIPTION:
Project Modifying Eating and Lifestyles at School (MEALS) was a school-based study developed by the nonprofit organization Project Bread (www.ProjectBread.org) and the Harvard School of Public Health. Project Bread hired a professional chef to work with several schools in a low-income, urban school district in Massachusetts to enhance the palatability and nutrient profile of the school meals. Four schools were randomly assigned to receive the professional chef. Additionally, two schools in that district and four schools in a second school district were randomly assigned to receive a behavioral psychology intervention to influence the selection and consumption of the healthier foods offered. Selection and consumption were assessed at baseline, up to 3 months post-implementation (short-term implementation for chef-enhanced meals), up to 4 months post-implementation (long-term implementation for behavioral psychology) and/or up to 7 months post-implementation (long-term implementation for chef-enhanced meals).

Primary Aim 1: to examine the impact of introducing healthier, chef-enhanced foods with increased palatability on selection and consumption among elementary and middle school students. It is hypothesized that there will be an increase in the selection and consumption of entrees, fruits, and vegetables in schools where healthier, chef-enhanced foods are served.

Aim 2: to examine the impact of physical modifications to the placement and displays of foods in the cafeteria on selection/consumption among elementary and middle school students. It is hypothesized that there will be an increase in selection and consumption of entrees, milk, fruits, and vegetables when modifications are made.

ELIGIBILITY:
Inclusion Criteria:

* Students in grades 1-8 attending a participating school and receiving a school meal on a study day

Exclusion Criteria:

* Bringing a lunch from home on a study day or not eating lunch in the cafeteria on a study day

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6873 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in the selection of meal components (Selection of entrees, milk, fruits, and vegetables) | baseline, up to 3 months post-implementation, and up to 7 months post-implementation
  Selection of entrees, milk, fruits, and vegetables
Change in the consumption of meal components (consumption of entrees, milk, fruits, and vegetables) | baseline, up to 3 months post-implementation, and up to 7 months post-implementation
  consumption of entrees, milk, fruits, and vegetables

SECONDARY OUTCOMES:
Time to eat (Estimated amount of time spent eating foods) | up to 24 months
  Estimated amount of time spent eating foods
Hunger (Self-reported hunger at the end of the meal) | up to 12 months
  Self-reported hunger at the end of the meal

REFERENCES:
- [Derived] Cohen JF, Richardson SA, Cluggish SA, Parker E, Catalano PJ, Rimm EB. Effects of choice architecture and chef-enhanced meals on the selection and consumption of healthier school foods: a randomized clinical trial. JAMA Pediatr. 2015 May;169(5):431-7. doi: 10.1001/jamapediatrics.2014.3805. PMID 25798990